CLINICAL TRIAL: NCT00059254
Title: Differential Metabolism of Dietary Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DMDFA (COMPLETED); R01DK055384 (NIH)
Record Dates: First submitted 2003-04-22; First posted 2003-04-23 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Diabetes; Hyperlipidemia
Keywords: fatty acids; oleic acid; palmitic acid; fat oxidation; energy expenditure; body composition; monounsaturated fat; human
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hyperlipidemias | interventions — Oleic Acid; Palmitic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oleic acid (OA) (Experimental)
  Interventions: Dietary Supplement: Oleic acid (OA)
- Palmitic acid (PA) (Experimental)
  Interventions: Dietary Supplement: Palmitic Acid (PA)

INTERVENTIONS:
Dietary Supplement: Oleic acid (OA) — OA-enriched (HI OA; fat, 40%; PA, 1.7%; OA, 31.4%)
  Arms: Oleic acid (OA)
Dietary Supplement: Palmitic Acid (PA) — PA-enriched (HI PA; fat, 40% of energy; PA, 16.8%; OA, 16.4%)
  Arms: Palmitic acid (PA)

SUMMARY:
Differences in how diet fats are converted to energy could explain some of the reported differences in health effects among different classes of dietary fat (e.g. monounsaturated vs. saturated). Recently, this laboratory showed that monounsaturated fats are turned into energy more readily than saturated fats. These results may mean that if one feeds more monounsaturated fatty acids (MUFA) and less saturated fatty acids (SFA) in the diet, body fat might accumulate at a lower rate. This could affect the risk of obesity and Type 2 Diabetes. This project has two principal Specific Aims which will be assessed in healthy young adults who are fed liquid formulas containing either an approximately equal amount of MUFA and SFA (controls) or a much greater amount of MUFA and much less SFA:

1. To determine if a higher intake of MUFA and a reciprocally lower intake of SFA is associated with a higher rate of fat oxidation. We hypothesize that the rate of fat oxidation after eating will be higher in those subjects randomized to the MUFA-enriched diet compared to controls.
2. To measure energy intake required to maintain constant body weight during each diet and to measure fat-free mass and fat mass, before and after each dietary change. We hypothesize that those on the high MUFA diet will need a higher energy intake required to maintain constant body weight.

DETAILED DESCRIPTION:
Our Preliminary Data indicate that the rate of oleic acid (OA) oxidation (amount/unit time) is 21% increased compared to palmitic acid (PA) when both fatty acids are fed to the same person at the same intake. We hypothesize that if the ratio of OA to PA in the diet were to increase, the rate of total fatty acid oxidation in the fed state also would increase under the same metabolic conditions. If our principal hypothesis is correct, overall daily fat balance might be decreased in humans fed diets enriched in OA. This would have potential significance to the treatment and prevention of obesity.

In order to address this hypothesis, we propose the following double-masked, randomized control trial. Indirect calorimetry will be performed in the fed and fasting state in young, healthy adults who will be studied under two conditions: after a 30-day, supervised, solid food diet and then again after a 30-day formula diet. The subjects will be randomized to receive either a Control Formula Diet of the same macronutrient and fatty acid composition as the solid food diet (OA=PA=16.4% total kcal) or a High Oleic Acid Formula Diet (OA=31.4% total kcal and PA=1.7% total kcal). The Control Diets (solid and liquid) provide amounts (per kcal) of total fat, saturated fat, and OA that are similar to the to the 50-75th percentile of intake of young adult Americans but above the intake of total fat and saturated fat that is recommended for optimal long-term health. The High OA Formula Diet is designed to simulate the fat source of the Mediterranean Diet. The High OA diet will result in a 167% increase in the intake/kcal of OA in the sn-1 and sn-3 positions of the dietary triacylglycerol. Using dual-energy x-ray absorptiometry (DEXA), we will monitor body composition before and after each diet, while adjusting energy intake to maintain constant body weight. The following Specific Aims will be addressed:

1. To determine if a higher intake of oleic acid (and a reciprocally lower intake of palmitic acid) is associated with a higher rate of fat oxidation. We hypothesize that the rate of fat oxidation (g/hr) in the fed state, adjusted for the covariate effect of the rate of fat oxidation on the solid food diet, will be higher (>30%) in those subjects randomized to the OA-enriched diet compared to controls. Furthermore, we hypothesize that fat oxidation will not be higher when expressed as a proportion of energy expenditure in the OA-enriched formula group. That is, we expect energy expenditure in the fed state to be higher in those fed the OA-enriched diet.
2. To measure energy intake required to maintain constant body weight during each diet and to measure fat-free mass and fat mass, before and after each dietary change. We hypothesize that a higher rate of fat oxidation on the high OA diet will be associated with a higher energy intake required to maintain constant body weight.
3. To compare fat oxidation on the liquid formula diet with that observed on the solid food diet. We hypothesize that fat oxidation will increase in those fed the OA-enriched diet.
4. To measure the thermic effect of feeding during both the solid food and formula diet periods. We hypothesize that the high OA feeding will be associated with a higher thermic effect of feeding.

ELIGIBILITY:
* Healthy young adults, ages 18-35 yr. .: Generally, this means that the subject is not being continually treated with medication (possible exceptions include thyroid replacement therapy and some allergy treatments).
* Must avoid pregnancy during the study duration (we will test for this as part of the protocol).
* Must avoid use of drugs that may affect lipid metabolism, including caffeine and nicotine.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2000-09 (Actual); Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Oxygen consumption | Day 29

SECONDARY OUTCOMES:
Carbon dioxide production | Day 29
Respiratory quotient | Day 29
excess Post exercise oxygen consumption (EPOC) | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Kein, MD, PhD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- Utmb Gcrc, Galveston, Texas, United States

REFERENCES:
- [Background] Schmidt DE, Allred JB, Kien CL. Fractional oxidation of chylomicron-derived oleate is greater than that of palmitate in healthy adults fed frequent small meals. J Lipid Res. 1999 Dec;40(12):2322-32. PMID 10588958
- [Result] Borsheim E, Kien CL, Pearl WM. Differential effects of dietary intake of palmitic acid and oleic acid on oxygen consumption during and after exercise. Metabolism. 2006 Sep;55(9):1215-21. doi: 10.1016/j.metabol.2006.05.005. PMID 16919541